CLINICAL TRIAL: NCT00001344
Title: Dextromethorphan Versus Placebo for Neuropathic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 930114; 93-D-0114
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-03

CONDITIONS: Diabetic Neuropathies; Herpes Zoster; Neuralgia
Keywords: Diabetes Mellitus; Diabetic Neuropathy; Memantine; NMDA Receptor Antagonists; Neuropathic Pain; Neuropathy; Post-Herpetic Neuralgia; Shingles
MeSH Terms: conditions — Diabetic Neuropathies; Herpes Zoster; Neuralgia; Diabetes Mellitus; Neuralgia, Postherpetic | interventions — Dextromethorphan

INTERVENTIONS:
Drug: dextromethorphan

SUMMARY:
In our current clinical trial, we are comparing the effects of two NMDA receptor antagonists to placebo in patients with painful distal symmetrical diabetic neuropathy or post-herpetic neuralgia. The treatments in this three-period crossover study are dextromethorphan, up to 920 mg/day (about 8 times the antitussive dose), memantine, 30-50 mg/day, and placebo. Memantine is an NMDA antagonist used in Europe to treat Parkinson's disease and Alzheimer's disease. The underlying hypothesis, based on studies of painful neuropathies in animal models, is that neuropathic pain is caused largely by sensitization of central nervous system neurons caused by excitatory amino acid neurotransmitters, acting largely through NMDA receptors. A previous small trial of dextromethorphan suggested efficacy in diabetic neuropathy pain. The study requires one visit to the NIH outpatient Pain Research Clinic, and consists of three 9-week treatment periods. Patients who respond to one of the medications will be invited to participate in further controlled studies of the medication followed by up to several years of open-label treatment under continued observation.

DETAILED DESCRIPTION:
In our current clinical trial, we are comparing the effects of two NMDA receptor antagonists to placebo in patients with painful distal symmetrical diabetic neuropathy or post-herpetic neuralgia. The treatments in this three-period crossover study are dextromethorphan, up to 920 mg/day (about 8 times the antitussive dose), memantine, 30-50 mg/day, and placebo. Memantine is an NMDA antagonist used in Europe to treat Parkinson's disease and Alzheimer's disease. The underlying hypothesis, based on studies of painful neuropathies in animal models, is that neuropathic pain is caused largely by sensitization of central nervous system neurons caused by excitatory amino acid neurotransmitters, acting largely through NMDA receptors. A previous small trial of dextromethorphan suggested efficacy in diabetic neuropathy pain. The study requires one visit to the NIH outpatient Pain Research Clinic, and consists of three 9-week treatment periods. Patients who respond to one of the medications will be invited to participate in further controlled studies of the medication followed by up to several years of open-label treatment under continued observation.

ELIGIBILITY:
Patients must be over 18 years of age.

Patients must have a definite diagnosis of diabetic neuropathy or post herpetic neuralgia or a diagnosis of neuropathic pain of various etiologies other than diabetic neuropathy or post herpetic neuralgia.

Duration of symptoms must be at least 3 months.

Severity of pain must be at least mild, if constant; or at least moderate, if intermittent and at least 2 hours duration a day.

Patients using tricyclics, narcotics, or antiseizure medications, must keep the drug dosages constant throughout the study.

No patients with unstable disease process; i.e., angina pectoris, accelerated hypertension, recent stroke or transient cerebral ischemia, uncontrolled seizures.

No pregnant or lactating women. Women of child bearing potential must use birth control pills, intrauterine device, or barrier contraceptive devices.

No history of significant drug abuse or PCP use. No history of IV drug abuse, prescription drug abuse, or alcoholism.

No significant liver or kidney disease.

No MAO inhibitors.

No cognitive impairment or language difficulty as judged by difficulty completing pain diary, medical history, or telephone conversation.

Patients must not have any other chronic pain condition that gives them pain greater than the neuropathy pain.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129
Dates: Start 1993-03; Study Completion 2001-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Albers GW, Saenz RE, Moses JA Jr, Choi DW. Safety and tolerance of oral dextromethorphan in patients at risk for brain ischemia. Stroke. 1991 Aug;22(8):1075-7. doi: 10.1161/01.str.22.8.1075. PMID 1866755
- [Background] Bakshi R, Faden AI. Competitive and non-competitive NMDA antagonists limit dynorphin A-induced rat hindlimb paralysis. Brain Res. 1990 Jan 15;507(1):1-5. doi: 10.1016/0006-8993(90)90512-a. PMID 1967971
- [Background] Choi DW. Dextrorphan and dextromethorphan attenuate glutamate neurotoxicity. Brain Res. 1987 Feb 17;403(2):333-6. doi: 10.1016/0006-8993(87)90070-9. PMID 2881608